CLINICAL TRIAL: NCT00753714
Title: Phase II, Randomised, Double-blind, Two-arm, Parallel Study of Vandetanib (ZACTIMA™ , ZD6474) Plus Gemcitabine (Gemzar® ) or Gemcitabine Plus Placebo as First Line Treatment of Advanced (Stage IIIB or IV) Non Small Cell Lung Cancer (NSCLC) Elderly Patients.
Brief Title: Zactima in Non Small Cell Lung Cancer (NSCLC) ELderly Patients In Combination With or Versus Gemcitabine
Acronym: ZELIG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4200L00012; EUDRACT n° 2007-004521-22
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: ZD6474; VANDETANIB; ZACTIMA; ADVANCED; NSCLC; LUNG CANCER; ELDERLY PATIENTS; GEMCITABINE; PHASE II; RANDOMIZED; DOUBLE-BLIND; histologically or cytologically-confirmed advanced (stage IIIB with supraclavicular lymph node metastases or pleural effusion or stage IV) NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Pleural Effusion | interventions — vandetanib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1.Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
  Interventions: Drug: ZD6474, Vandetanib; Drug: Gemcitabine
- B (Placebo Comparator): Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1.Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with placebo alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
  Interventions: Drug: Placebo to Match ZD6474, Vandetanib; Drug: Gemcitabine

INTERVENTIONS:
Drug: ZD6474, Vandetanib — 100 mg as a once daily oral dose, from Day 1 until disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Zactima
  Arms: A
Drug: Placebo to Match ZD6474, Vandetanib — 100 mg as a once daily oral dose, from Day 1 UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Zactima
  Arms: B
Drug: Gemcitabine — administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle UP to 6 cycles or UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Gemzar

SUMMARY:
The primary objective of this study is to demonstrate an improvement in Progression-Free Survival (PFS) for the combination of vandetanib plus gemcitabine compared with gemcitabine plus placebo in chemonaïve (not including an adjuvant regimen) patients aged ≥ 70 years with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of advanced NSCLC (stage IIIB with supraclavicular lymph node metastases or pleural effusion or stage IV) on entry into study
* One or more measurable lesions at least 10 mm in the longest diameter (LD) by spiral CT scan or 20 mm with conventional techniques according to RECIST criteria
* Chemotherapy-naïve (prior chemotherapy in the adjuvant setting completed more than 3 months before the trial entry is accepted).
* Female or male aged 70 years or above

Exclusion Criteria:

* Patients must not have received prior anti-cancer therapy except in the adjuvant setting
* Inadequate end-organ function or Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial
* Significant cardiovascular event (e.g. myocardial infarction, superior vena cava [SVC] syndrome, New York Heart Association [NYHA] classification of heart disease ³2) within 3 months before entry, or presence of cardiac disease that in the opinion of
* History of arrhythmia or QTc with Bazett's correction unmeasurable or ≥ 480 msec on screening ECG

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Italy (15):
  - Research Site, Meldola, (fc)
  - Research Site, Avellino, AV
  - Research Site, Bari, BA
  - Research Site, Treviglio, BG
  - Research Site, Bologna, BO
  - Research Site, Genova, GE
  - Research Site, Taormina, ME
  - Research Site, Milan, MI
  - Research Site, Perugia, PG
  - Research Site, Ravenna, RA
  - Research Site, Roma, Roma
  - Research Site, Trento, TN
  - Research Site, Orbassano, TO
  - Research Site, Udine, UD
  - Research Site, Padua

REFERENCES:
- [Background] Gridelli C. Treatment of advanced non small-cell lung cancer in the elderly: from best supportive care to the combination of platin-based chemotherapy and targeted therapies. J Clin Oncol. 2008 Jan 1;26(1):13-5. doi: 10.1200/JCO.2007.14.1820. No abstract available. PMID 18165633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 124 patients have been enrolled in a period of 19 months in 17 actively recruiting Oncologic Medical Department in Italy.
Groups:
- ZD6474 (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1. Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
- Placebo to Match ZD6474 (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1. Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with placebo alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued
Period: Overall Study
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Started | 61 | 63
Completed | 1 | 1
Not Completed | 60 | 62
Not completed — Lack of Efficacy | 21 | 34
Not completed — Adverse Event | 26 | 18
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 3 | 3
Not completed — Other | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- ZD6474 (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1. . Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
- Placebo to Match ZD6474 (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1. . Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with placebo alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
- Total: Total of all reporting groups
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.03 (3.34) | 75.48 (3.49) | 75.25 (3.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: Oct 2008- dec 2011
Measure: Median (95% Confidence Interval); unit: days
Groups:
- ZD6474 (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1.Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Number analyzed (Participants) | 61 | 63
days | 183 [116 to 214] | 169 [95 to 194]

2. Secondary Outcome: Overall Survival
Time Frame: Oct 2008- dec 2011
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Number analyzed (Participants) | 61 | 63
days | 262 [170 to 356] | 305 [214 to 355]

3. Secondary Outcome: Overall Objective Response
Time Frame: Oct 2008- dec 2011
Measure: Number; unit: Participants
Groups:
- ZD6474 ( (Vandetanib),Gemcitabine: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1. . Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
Arm/Group | ZD6474 ( (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Number analyzed (Participants) | 61 | 63
Participants | 9 | 8

4. Secondary Outcome: Duration of Response
Time Frame: Oct 2008- dec 2011
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Number analyzed (Participants) | 61 | 63
days | 225 [175 to NA] — Too few participants experienced event to compute upper limit of CI, i.e.sample analyzed is to small compared with the initial statistical plan or when less than 50% of the subjects are available for analysis | 214 [124 to 232]

5. Secondary Outcome: The Safety and Tolerability Profile of ZD6474 (Vandetanib) in Combination With Gemcitabine
Description: The Safety and Tolerability Profile of ZD6474 (Vandetanib) in Combination With Gemcitabine is defined as the number of Adverse Events which includes any symptoms and/or Clinically Significant Laboratory or Vital Signs Abnormalities, and/or ECGs Changes
Time Frame: Oct 2008- Dec 2011
Measure: Number; unit: Adverse Events
Arm/Group | ZD6474 (Vandetanib),Gemcitabine | Placebo to Match ZD6474 (Vandetanib),Gemcitabine
Number analyzed (Participants) | 61 | 63
Adverse Events | 378 | 381

ADVERSE EVENTS:
Groups:
- ZD6474 (Gemcitabine), Vandetanib: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1. . Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with vandetanib alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued.
- Placebo to Match ZD6474 (Gemcitabine), Vandetanib: Gemcitabine administered intravenously at 1200 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1. . Patients will receive gemcitabine for up to a maximum of 6 cycles, after which period patients should continue on daily oral dosing with placebo alone until progression. Once a patient has met the study criteria for disease progression on vandetanib/gemcitabine or placebo/gemcitabine, randomised treatment must be permanently discontinued
Arm/Group | ZD6474 (Gemcitabine), Vandetanib | Placebo to Match ZD6474 (Gemcitabine), Vandetanib
Serious Adverse Events (participants affected / at risk) | 26/61 | 25/63
Other Adverse Events (participants affected / at risk) | 59/61 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 (Gemcitabine), Vandetanib (N=61) | Placebo to Match ZD6474 (Gemcitabine), Vandetanib (N=63)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Pulmunary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmunary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
acute pulmunary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
chronic obstructive pulmunary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
tachycardia (Cardiac disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Depressed Level Of Consciuosness (Nervous system disorders) | 1 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 2 | 0
Uraniry Retention (Renal and urinary disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Eye Disorder (Eye disorders) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight Decrease (Investigations) | 1 | 0
Muscoloskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ear Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 3
Chest Pain (General disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 (Gemcitabine), Vandetanib (N=61) | Placebo to Match ZD6474 (Gemcitabine), Vandetanib (N=63)
pyrexia (General disorders) | 17 | 17
Fatigue (General disorders) | 14 | 15
Asthenia (General disorders) | 9 | 13
Dispnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10
PLT count decrease (Blood and lymphatic system disorders) | 7 | 9
Neutropenia (Blood and lymphatic system disorders) | 12 | 12
Anaemia (Blood and lymphatic system disorders) | 8 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 9 | 9
Nausea (Gastrointestinal disorders) | 7 | 8
Vomiting (Gastrointestinal disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 15 | 5
Anorexia (Metabolism and nutrition disorders) | 8 | 17
Hypokaliemia (Metabolism and nutrition disorders) | 2 | 7
Mucosal Inflammation (General disorders) | 4 | 4
Oedema Peripheral (General disorders) | 4 | 12
Chest Pain (General disorders) | 2 | 15
Pulmunary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Alanine Aminotransferase Increased (Blood and lymphatic system disorders) | 5 | 1
Neutrphil Count Decreased (Blood and lymphatic system disorders) | 5 | 2
Aspartate Aminotransferase Inctìreased (Blood and lymphatic system disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Phlebitis (Vascular disorders) | 5 | 3
Depression (Psychiatric disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.